CLINICAL TRIAL: NCT06222203
Title: Surveillance for Malignant Transformation of Neurofibromatosis Type 1 (NF1) Related Peripheral Nerve Sheath Tumors (PNST)
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001696; 001696-C
Record Dates: First submitted 2024-01-23; First posted 2024-01-24 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09-24

CONDITIONS: Neurofibromatosis 1; Nerve Sheath Neoplasms
Keywords: NF1; atypical neurofibromas; Plexiform Neurofibromas; neurofibromas; PN; MPNST; malignant transformation; distinct nodular lesion
MeSH Terms: conditions — Neurofibromatosis 1; Nerve Sheath Neoplasms; Neurofibroma, Plexiform; Neurofibroma; Neurofibrosarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1 - High-Risk: Participants with clinical or genetic diagnosis of NF1 AND at least one of the eligibility-required high-risk characteristics
- 2 - Low-Risk: Participants with clinical or genetic diagnosis of NF1 AND none of the eligibility-required high-risk characteristic
- 3 - Caregiver: Parents or guardians of participants 8-17 years old in High-Risk or Low-Risk Cohorts

SUMMARY:
Background:

Neurofibromatosis type 1 (NF1) is a genetic disease that can cause many symptoms. About half of people with NF1 will develop benign (noncancerous) tumors along nerves in the skin, brain, and other parts of the body. Sometimes, though, these tumors can become cancerous. Researchers do not yet know how to predict which tumors will become cancerous.

Objective:

To test a new method for predicting which benign NF1 tumors will become cancerous.

Eligibility:

People aged 3 years and older with a clinical or genetic diagnosis of NF1.

Design:

* Participants will be screened with a review of their medical history. All participants will have a baseline visit. They will have bood tests and imaging scans. They will have a physical exam. They will answer questions about their family history. Participants aged 8 years and older will take tests of their thinking skills and their emotional health.
* Some participants may be asked to undergo more tests. These may include another type of imaging scan and a biopsy: A small sample of tissue may be removed from the tumor.
* Participants will be divided into two groups: those believed to be at low risk and those believed to be at high risk of developing cancer.
* Participants in the high-risk group will be asked to return for their next visit in 1 month to 3 years.
* Participants in the low-risk group will be asked to return for their next visit in 6 months to 5 years.
* Participants may also have follow-up visits by phone throughout the study. They will be in the study for 10 years.

DETAILED DESCRIPTION:
Background

* Patients with NF1 are at risk for the development of both benign and malignant peripheral nerve sheath tumors (MPNST). Some factors that increase risk for malignant tumors are known, such as large benign plexiform neurofibroma (PN) tumor burden, germline NF1 microdeletion, and history of radiation therapy. However, there is not currently a consensus in the field about the most appropriate clinical surveillance or management strategy for these patients at increased risk of malignancy.
* In the past decade, data from the existing NCI POB NF1 Natural History study (08-C-0079, NCT00924196) and others have identified atypical neurofibromas (AN) and atypical neurofibromatous neoplasms of uncertainly biologic potential (ANNUBP) as premalignant lesions characterized by heterozygous loss of CDKN2A/B in addition to the homozygous loss of NF1 found in all PN.
* On Magnetic Resonance Imaging (MRI), distinct nodular lesions (DNL) have been identified as having unique characteristics, including increased fluorodeoxyglucose (FDG)-positron emission tomography (PET) avidity and growth rate compared to surrounding PN, and are often, though not always, found to be AN on histologic evaluation.

Objective

- To assess the feasibility of the study algorithm in identifying ANs, ANNUBPs, CDKN2A/B mutated lesions, and/or MPNST

Eligibility

* Participants aged >= 3 years old with a clinical or genetic diagnosis of NF1.
* Participants will be enrolled in one of the following cohorts:

  * For the High-Risk Cohort one of the following criteria: microdeletion or 844-848 missense variants or other variants associated with increased risk of MPNST, family history of MPNST/ANNUBP/AN, personal history of MPNST/ANNUBP/AN or neurofibroma with CDKN2A/B loss, prior radiation therapy at any site, large PN burden (>= 350 mL), or presence >= 1 DNL at baseline.
  * For the Low-Risk Cohort: none of the criteria noted for the high-risk cohort beyond NF1 diagnosis.

Design

* This is an observational study to identify risk factors associated with severe disease in NF1 and to assess the feasibility of a novel NF1 Increased MPNST Risk Surveillance and Management Algorithm to aid in the surveillance and management of participants with NF1.
* 225 participants will be enrolled in this study.

ELIGIBILITY:
* INCLUSION CRITERIA:

High-Risk and Low-Risk NF1 Cohorts

* Age >= 3 years old
* Participants with clinical or genetic diagnosis of NF1.
* Participants with a diagnosis of mosaic or segmental NF1 are also eligible.
* Individuals may have (High-Risk Cohort) or not have (Low-Risk Cohort) at least one of the following characteristics:

  * Microdeletion or 844-848 missense variants or other variants associated with increased risk of malignant peripheral nervous sheath tumor (MPNST)
  * Family history of MPNST / atypical neurofibromatous neoplasm of unknown biologic potential (ANNUBP) / atypical neurofibromas (ANF)
  * Personal history of MPNST/ANNUBP/ANF or neurofibroma with CDKN2A loss
  * Prior radiation therapy at any site
  * Large plexiform neurofibroma (PN) burden (>= 350 mL)
  * Presence >= 1 DNL at baseline
* The ability of the individual, parent/guardian or Legally Authorized Representative (LAR) to understand and the willingness to sign a written consent document for participation.

EXCLUSION CRITERIA:

High-Risk and Low-Risk NF1 Cohorts

- Inability or unwillingness to undergo MRI imaging

INCLUSION CRITERIA:

Parent Cohort

* Parent or guardian of pediatric individuals (8-17 years old) in High-Risk or Low-Risk Cohorts.
* The ability of the parent/guardian or LAR to understand and the willingness to sign a written consent document for parent/guardian participation in this study.

EXCLUSION CRITERIA:

Parent Cohort

- None.

Ages: 3 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants aged >= 3 years old with a clinical or genetic diagnosis of NF1; parents or guardians of participants ages 8-17 years old.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Assess feasibility of the study algorithm in identifying atypical neurofibromas (ANs), atypical neurofibromatous neoplasms of unknown biologic potential (ANNUBPs), CDKN2A/B mutated lesions, and/or malignant peripheral nervous sheath tumors (MPNS... | Throughout the study
  Proportion of lesions that undergo surgical intervention (biopsy or resection) that are ANs, ANNUBPs, CDKN2A mutated lesions and/or MPNST

SECONDARY OUTCOMES:
Assess whether the proposed surveillance and management approach for participants with NF1 at high risk and low risk of MPNST is feasible | Throughout the study
  Number of participants complying with recommendations for imaging/surgical interventionsNumber of resections recommended vs successfully completedProportion of subjects from the low-risk cohort that transition to the high- risk algorithm during the study observation periodThe number of subjects who develop high grade MPNST during the observation periodNumber of subjects who develop high grade MPNST outside of a pre-existing DNL or PN during the observation periodData from the Tumor Specific Risk Factor and Participant Specific Risk Factor Checklists

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte C Widemann, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP
Time Frame: Data from this study may be requested from other researchers after the completion of the primary endpoint. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Data from this study may be requested by contacting the PI. Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001696-C.html